CLINICAL TRIAL: NCT04399759
Title: Investigation of the Effect on Instrumental Activities of Daily Living Approach in Home Environment for Patients With Stroke
Brief Title: Instrumental Activities of Daily Living Approach in Home Environment for Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, En-Chi Chiu, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CTH-108-2-5-029
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Stroke; Activities of Daily Living
Keywords: Stroke; Activities of Daily Living; Home Care Services
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-IADL Group (Experimental): Approach-Instrumental Activities of Daily Living in home
  Interventions: Behavioral: Approach-Instrumental Activities of Daily Living
- Control group (Active Comparator): Home health education
  Interventions: Behavioral: Home health education

INTERVENTIONS:
Behavioral: Approach-Instrumental Activities of Daily Living — Individualized instrumental activities of daily living training
  Arms: A-IADL Group
Behavioral: Home health education — Individualized home health education
  Arms: Control group

SUMMARY:
The purpose of this study was to conduct a randomized clinical trial. Implement instrumental daily activities of daily living (A-IADL) in home rehabilitation. To explore the effect of A-IADL on stroke patients' movement, cognition, social participation, daily life function and quality of life.

DETAILED DESCRIPTION:
Subjects were randomized to intervention group and control group. The experiment was designed as randomized cross-over control trial. The primary outcome included 11 measures, Fugl-Meyer Assessment, Balance computerized adaptive testing, Mini Mental State Examination, Participation Measure-3 Domains ,4 Dimensions, Canadian Occupational Performance Measure, Barthel Index-based Supplementary Scales, Frenchay Activities Index, Lawnton Instrumental Activities of Daily Living, stroke impact scale, Stroke Self-Efficacy Questionnaire, and Kingston Caregiver Stress Scale.

ELIGIBILITY:
Inclusion Criteria:

* age > 20 years
* Diagnosis of stroke
* The modified Rankin Scale : 2~4
* Keep sitting for half an hour by himself/herself
* Follow instructions
* Willing to sign the subject's consent

Exclusion Criteria:

* Diagnosis of dementia
* History of orthopedic diseases or peripheral nerve injury

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | Baseline to 6 weeks
  The Fugl-Meyer Assessment scale is an index to assess the sensorimotor impairment in individuals who have had stroke. The score ranges is 0 to 226. A higher score indicates better body function.
Balance computerized adaptive testing | Baseline to 6 weeks
  The Balance computerized adaptive testing is a test about stroke patients, includes movement, balance, activities of daily living.
Mini Mental State Examination | Baseline to 6 weeks
  The Mini Mental State Examination general cognitive function. The score ranges is 0 to 30. A higher score indicates better general cognitive function.
Participation Measure-3 Domains ,4 Dimensions | Baseline to 6 weeks
  The Participation Measure-3 Domains, 4 Dimensions assesses social participation. A higher score indicates better social participation.
Canadian Occupational Performance Measure | Baseline to 6 weeks
  The COPM protocol is divided into three areas: self-care, productivity, and leisure. Patients define important activities and classify them with a score of one to 10. A higher score indicates better occupational performance.
Barthel Index (BI) -based Supplementary Scales | Baseline to 6 weeks
  The Barthel Index-based Supplementary Scales assesses basic activities of daily living using three scales:actual performance, ability, and self-perceived difficulty. The score ranges the three scales (i.e., actual performance, ability, and self-perceived difficulty)is 0-20, 0-18, and 0-20, respectively. A higher score indicates better basic activities of daily living.
Frenchay Activities Index | Baseline to 6 weeks
  The Frenchay Activities Index is a measure of instrumental activities of daily living for use with patients recovering from stroke. The score ranges is 0 to 45. A higher score indicates better instrumental activities of daily living.
Lawnton Instrumental Activities of Daily Living | Baseline to 6 weeks
  The Lawnton Instrumental Activities of Daily Living assesses instrumental activities of daily living.The score ranges is 0 to 8. A higher score indicates better instrumental activities of daily living.
Stroke Impact Scale | Baseline to 6 weeks
  The Stroke Impact Scale assesses other dimensions of health-related quality of life: emotion, communication, memory and thinking, and social role function.The score ranges is 59 to 295. A lower score indicates the quality of life less affected by stroke.
Stroke Self-Efficacy Questionnaire | Baseline to 6 weeks
  The Stroke Self-Efficacy Questionnaire is a self-report scale measuring self-efficacy judgments in specific domains of functioning post stroke. The score ranges is 0 to 130. A higher score indicates better self-efficacy.
Kingston Caregiver Stress Scale | Baseline to 6 weeks
  The Kingston Caregiver Stress Scale is a self-report scale measuring caregiver stress. The score ranges is 10 to 50. A higher score indicates greater stress.

CONTACTS AND LOCATIONS:
Overall Officials: En-Chi Chiu, PhD, Study Director — National Taipei University of Nursing and Health Sciences
Locations (1):
- Cardinal Tien Hospital, New Taipei City, Xindian Dist, Taiwan

REFERENCES:
- [Derived] Gibson E, Koh CL, Eames S, Bennett S, Scott AM, Hoffmann TC. Occupational therapy for cognitive impairment in stroke patients. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD006430. doi: 10.1002/14651858.CD006430.pub3. PMID 35349186